CLINICAL TRIAL: NCT03207633
Title: Comparative Study of the Therapeutic Effect of Low Frequency TMS on DLPFC and OFC in OCD Patients
Brief Title: Low Frequency TMS on DLPFC and OFC in OCD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professorf, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Low frequency TMS in OCD
Record Dates: First submitted 2017-06-24; First posted 2017-07-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Psychiatric Disorder
Keywords: OCD, rTMS, right orbitofrontal cortex
MeSH Terms: conditions — Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First group (Active Comparator): First group (20 patients) receive for 10 sessions of low frequency rTMS targeting right DLPFC by means of a Butterfly coil using the following parameters: 120% RMT, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool.
  Interventions: Procedure: Repetitive trans-magnetic stimulation (rTMS) on DLPFC
- Second group (Active Comparator): The second group (20 patients) will receive 10 sessions of low-frequency rTMS over the right orbitofrontal cortex (OFC) by means of a Butterfly coil using the following parameters: 120% motor threshold, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool.
  Interventions: Procedure: Repetitive trans-magnetic stimulation (rTMS) on OFC
- Third group (Sham Comparator): The third group (the sham condition) (20 patients) will receive sham stimulations of rTMS with the same pulse delivery as the other groups but with the coil placed perpendicular to the scalp.
  Interventions: Procedure: Sham repetitive trans-magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive trans-magnetic stimulation (rTMS) on DLPFC — Repetitive trans-magnetic stimulation (rTMS) on DLPFC
  Arms: First group
Procedure: Repetitive trans-magnetic stimulation (rTMS) on OFC — Repetitive trans-magnetic stimulation (rTMS) on OFC
  Arms: Second group
Procedure: Sham repetitive trans-magnetic stimulation (rTMS) — Sham repetitive trans-magnetic stimulation (rTMS)
  Arms: Third group

SUMMARY:
This study aims to evaluate the therapeutic effect of low frequency rTMS over the right DLPFC, versus right OFC versus Sham group of obsessive-compulsive disorder (OCD) patients. Sixty patients will be recruited from the out-patient psychiatric clinic of a university hospital, and randomized into three equal groups. The 1st group will receive 10 sessions of low frequency rTMS targeting right DLPFC by means of a butterfly coil, 120% RMT, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool. The 2nd group will receive 10 sessions of low-frequency rTMS over the right orbitofrontal cortex (OFC), the international 10-20 EEG system will be used to position the coil over the right OFC, at the right frontopolar 2 (Fp2) electrode site, using the following parameters: 120% motor threshold, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool. The 3rd group will receive sham stimulations with the same pulse delivery as the other groups but with the coil placed perpendicular to the scalp.

The resting motor threshold (RMT) and cortical silent period (CSP) at different intensities from 110 % to 150 % will be measured before and after the end of sessions. All assessments like (Y-BOCS), (HAM-A), Beck Depression Inventory, (CGI-S), (MoCA) will be performed before and after end of the sessions and 3 months later.

DETAILED DESCRIPTION:
This study aims to evaluate the therapeutic effect of low frequency rTMS over the right DLPFC, versus right OFC versus Sham group of OCD patients. Sixty patients will be recruited from the out-patient psychiatric clinic of a university hospital, the patients will be randomized into three groups (20 patients for each group) using closed envelopes.

The first group (20 patients) will receive 10 sessions of low frequency rTMS targeting right DLPFC by means of a Butterfly coil, The DLPFC stimulation site was defined as the region 5 cm dorsolateral in the same sagittal plane as the optimal site for MT production in the first dorsal interosseous, using the following parameters: 120% RMT, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool.

The second group (20 patients) will receive 10 sessions of low-frequency rTMS over the right orbitofrontal cortex (OFC) by means of a butterfly coil, the international 10-20 EEG system will be used to position the coil over the right OFC, at the right frontopolar 2 (Fp2) electrode site, using the following parameters: 120% motor threshold, 1 Hz, 3 trains, each of 500 pulses with a 40 seconds inter-train interval allowing the coil to cool.

The third group (the sham condition) (20 patients) group will receive sham stimulations with the same pulse delivery as the other groups but with the coil placed perpendicular to the scalp.

The resting motor threshold (RMT) and cortical silent period (CSP) at different intensities from 110 % to 150 % will be measured before and after the end of sessions. All assessments like (Y-BOCS), (HAM-A), Beck Depression Inventory, (CGI-S), (MoCA) will be performed before and after end of the sessions and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* being 18 or over
* being assigned a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) or DSM-V diagnosis of OCD by the referring psychiatrist

Exclusion Criteria:

* (1) presenting established cognitive or communication problems which makes it challenging to understand the questionnaires and take part in the therapeutic encounters
* (2) suffering from other severe psychiatric disorders, metabolic, or neurological disorders .
* (3) Patients with pacemaker, or metallic devices

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Three months
  Assessment of Obsessive Compulsive disorder using (Y-BOCS)
Hamilton Anxiety Rating Scale (HAM-A) | Three months
  Assessment of anxiety using Hamilton scale
Beck Depression Inventory | Three months
  Assessment of Depression using Beck depression inventory
Clinical Global Impression-Severity scale (CGI-S) | Three months
  Assessment of clinical severity using CGI-S
Montreal Cognitive Assessment (MoCA) | Three months
  Assessment of cognitive function using (MoCA)

SECONDARY OUTCOMES:
Changes of cortical excitability parameters (RMT and CSP) | Ten days
  Measurment of changes of cortical excitability parameters (RMT and CSP) before and after sessions in the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Khedr, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University
Locations (1):
- Eman Khedr, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No